CLINICAL TRIAL: NCT06700083
Title: Safety, Tolerability, and Pharmacokinetics of Single and Multiple Subcutaneous Injections of SHR-6934 in Healthy Subjects: a Randomized, Double-blind, Dose-escalation, Placebo-controlled Phase I Trial
Brief Title: A Safety, Tolerability, Pharmacokinetic Study of SHR-6934 Injection in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-6934-101
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- SAD dose 1 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- SAD dose 2 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- SAD dose 3 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- SAD dose 4 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- SAD dose 5 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- SAD dose 6 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- MAD dose 1 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- MAD dose 2 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- MAD dose 3 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo
- MAD dose 4 (Experimental)
  Interventions: Drug: SHR-6934 injection; Drug: SHR-6934 placebo

INTERVENTIONS:
Drug: SHR-6934 injection — SHR-6934 injection
Drug: SHR-6934 placebo — SHR-6934 placebo

SUMMARY:
This study was a randomized, double-blind, single-dose and multi-dose, placebo-controlled phase Ⅰ clinical trial. Six dose groups were planned for the SAD part of the study and four dose groups were planned for the MAD part. A total of 88 healthy subjects were included.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and methods, voluntarily participate in the study, comply with study requirements, and sign the written informed consent form (ICF);
2. Male or female aged 18-60;
3. Females must have a negative pregnancy test at the Screening Visit;
4. Body mass index (BMI) between 19 and 28 kg/m2;
5. Normal Electrocardiogram (ECG);
6. Men and women of childbearing potential must agree to take effective contraceptive methods.

Exclusion Criteria:

1. History of any clinically important disease or disorder;
2. History of drug or other allergies, or who, in the judgement of the investigator, may be allergic to the study drug or any component of the study drug;
3. Prior history of risk factors for Torsades de Pointes, such as unexplained syncope, definite long QT syndrome (including family history), heart failure, myocardial infarction, angina pectoris;
4. Systolic blood pressure (SBP)≥140 mmHg or <90 mmHg, diastolic blood pressure (DBP) ≥90 mmHg or <60 mmHg;
5. Patients with orthostatic hypotension;
6. Positive results of hepatitis B surface antigen, hepatitis C antibody, syphilis antibody and human immunodeficiency virus antibody.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of subjects with adverse events (AEs) | Baseline up to 113 days after the last dosing

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration (AUC0-t) for SHR-6934 | Baseline up to 113 days after the last dosing
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞) for SHR-6934 | Baseline up to 113 days after the last dosing
Maximum plasma concentration (Cmax) for SHR-6934 | Baseline up to 113 days after the last dosing
Time to reach maximum plasma concentration (Tmax) for SHR-6934 | Baseline up to 113 days after the last dosing
Terminal half-life (t1/2) for SHR-6934 | Baseline up to 113 days after the last dosing
Apparent clearance (CL/F) of SHR-6934 for administration subcutaneously | Baseline up to 113 days after the last dosing
Apparent volume of distribution (V/F) of SHR-6934 for administration subcutaneously | Baseline up to 113 days after the last dosing
Proportion of anti-drug antibodies (ADA) positive subjects | Baseline up to 113 days after the last dosing
Baseline and placebo-adjusted QTcF after SHR-6934 | Baseline up to 15 days after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided